CLINICAL TRIAL: NCT00469508
Title: A Randomized, Double-Blind, Placebo-Controlled Evaluation of Modafinil vs Placebo for the Treatment of Methamphetamine Dependence
Brief Title: Modafinil vs Placebo for the Treatment of Methamphetamine Dependence
Acronym: Modafinil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steve Shoptaw, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P50DA018185-03 (NIH); P50DA018185 (NIH); NCT00462293 (obsolete NCT alias)
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Methamphetamine Dependence
Keywords: Methamphetamine; Modafinil; Medication; Contingency Management; Crystal meth; Los Angeles; Addiction; Meth
MeSH Terms: conditions — Behavior, Addictive | interventions — Modafinil; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modafinil (Active Comparator): Modafinil 400mg oral dose taken daily for 12 weeks
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): Modafinil 0mg (sugar pill) oral dose taken daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — 400mg pills taken orally daily for 12 wks.
  Other Names: Provigil
  Arms: Modafinil
Drug: Placebo — 400mg pills taken orally daily for 12 wks
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Modafinil is a non-amphetamine type stimulant that acts as a wakefulness-promoting drug, and is approved for managing symptoms of narcolepsy (i.e., daytime somnolence). Its precise mechanism of action in promoting wakefulness remains unclear. This trial is a placebo-controlled double-blind trial of modafinil, on a platform of contingency management (CM) and individual cognitive-behavioral (CBT) counseling, for the treatment of methamphetamine dependence. Participants in this study will complete a 2-week baseline screening period during which they will provide urine samples and complete physical and psychological assessments to establish their eligibility for the study. In addition, participants will be asked to provide a blood or saliva specimen for genetic testing in order to identify genetic variations that influence response to methamphetamine and to treatment with modafinil. Upon successful completion of screening, participants will be randomly assigned to receive either modafinil (400mg qd) or placebo during the 12 weeks of the study. Neither the participants nor study staff will know who is receiving active medication or placebo. Regardless of medication condition, all participants will receive CM and weekly individual CBT counseling sessions to help them stop using methamphetamine and prevent relapse. They will attend the clinical research site (either at the UCLA Hollywood Clinic, or the Rancho Cucamonga site) three times per week, providing urine samples at each visit, completing data measures, and receiving individual CBT counseling on one visit each week. At the end of the 12-week study, the medication or placebo will be discontinued. Participants will return to the research site approximately 30 days following medication discontinuation for a brief health check to assess any possible lingering side effects and complete brief data measures.

DETAILED DESCRIPTION:
This application proposes a placebo-controlled double-blind trial of modafinil, on a platform of contingency management (CM) and individual cognitive-behavioral counseling (CBT once weekly individual session), for the treatment of methamphetamine dependence. Modafinil is a medication warranting evaluation as a treatment for MA dependence. It has a half-life of approximately 15 hours and reaches steady state in 2-4 days (Package insert) and will likely require once daily dosing, which reduces problems with medication adherence. Modafinil has potent psychiatric and behavioral effects that include brightening mood (Menza et al., 2000; Ninan et al., 2004), improving cognition (Turner et al., 2004a, b; 2003), improving impulse control (Turner et al., 2003; Turner et al., 2004a), and countering fatigue (Beusterien et al., 1999, Stahl et al., 2003). These effects neatly counterbalance effects produced by MA withdrawal (Newton et al., 2004) and may have particular value in ameliorating the negative reinforcing properties of MA, i.e., when MA is used to immediately relieve depressed mood due to recent abstinence (Peck et al., 2005b). CM is a behavioral intervention that effectively helps substance abusers to initiate abstinence, particularly from cocaine (Higgins et al., 1993; Higgins et al., 2000; Higgins et al., 1991) and from methamphetamine (Roll & Shoptaw, in press; Shoptaw et al., 2005). As well, CM has been shown to reduce substance abuse and optimize the effects of medications in reducing substance abuse (Carroll, 2004; Shoptaw et al., 2002). The objective of this study is to determine whether modafinil reduces methamphetamine use and concomitant physical and psychological symptoms more effectively than placebo when administered in conjunction with CM and CBT. The purpose of this project is to evaluate whether methamphetamine abusers seeking outpatient treatment demonstrate significantly significant reductions of methamphetamine when randomly assigned to receive modafinil (400mg qd) in combination with CM and weekly CBT compared their peers randomly assigned to receive placebo in combination with CM and weekly CBT.

Research Hypotheses:

1. Participants receiving active experimental drug (modafinil 400mg) will demonstrate statistically significant reductions in methamphetamine use over participants receiving placebo. Methamphetamine use outcomes will be measured using urine samples and analyzed with the following indices: Treatment Effectiveness Score, the Joint Probability Index, self-report of methamphetamine use verified by urine drug screening, and the longest uninterrupted period of methamphetamine abstinence. Primary analyses will be conducted using modeling approaches (Generalized Estimation Equations, Markov Chain Transition Models) depending upon the structure of the dataset. Self-report of methamphetamine use will be analyzed using the Addiction Severity Index drug composite scale and Substance Use Inventory (SUI).
2. Participants receiving active experimental drug will remain in treatment for significantly longer periods compared to participants receiving placebo. Retention will be measured by the number of days in the protocol and analyzed using survival analysis.

   a. Specifically, participants with mild cognitive dysfunction (as measured as <=1 SD below the published mean for the MicroCog assessments) receiving modafinil (400mg) will demonstrate significantly greater overall retention, and attendance to CBT sessions than those participants with cognitive function measured at greater than 1 SD below the mean for the MicroCog assessments who are receiving placebo.
3. Participants receiving active experimental drug (modafinil 400mg) will demonstrate statistically significant reductions in reported methamphetamine craving over participants receiving placebo. Craving outcomes will be measured using a visual analogue scale.
4. Participants receiving active experimental drug (modafinil 400mg) will demonstrate statistically significant reductions in withdrawal symptoms and somatic complaints compared to participants receiving placebo. These outcomes will be measured using the BSI, the Beck Depression Inventory-II, and the Quality of Well-Being scale.

Exploratory analyses will also be conducted to identify potential genetic variants associated with treatment response to modafinil for MA dependence. Candidate genes implicated by previous research as being involved in the pathogenesis of MA dependence and/or the molecular mechanism of modafinil (for example, genes for neurotransmitter receptors and transporters, including dopamine, norepinephrine, GABA, and glutamate, as well as genes for enzymes involved in the metabolism of these neurotransmitter, such as catechol-O-methyltransferase and monoamine oxidase A) will be sequenced in order to determine the frequency of known single nucleotide polymorphisms (SNPs), as well as potentially identify novel SNPs, in these genes among MA dependent participants. Initial analyses will focus on genes involved in the dopaminergic pathway, given the importance of dopamine in the neurobiology of MA dependence, but additional genes may also be assessed. SNPs associated with response to modafinil will be identified in order to generate hypotheses for future pharmacogenomic studies.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. meet DSM-IV criteria for methamphetamine dependence;
3. willing and able to comply with study procedures;
4. willing and able to provide written informed consent;
5. if female, not pregnant or lactating and willing to use an acceptable method of barrier birth control (e.g. condoms) during the trial and for one month after discontinuation of study medication (modafinil may reduce the effectiveness of steroidal contraceptives both during administration and for one month after discontinuation).

Exclusion Criteria:

1. have a medical condition that, in the study physician's judgment, may interfere with safe study participation (e.g., active TB, unstable cardiac, renal, or liver disease, unstable diabetes, or elevated liver enzymes (SGOT or SGPT) greater than 4 times the upper limit of normal);
2. have a current neurological disorder (e.g., organic brain disease, dementia) or major psychiatric disorder not due to substance abuse (e.g., schizophrenia or bipolar illness) as assessed by the SCID and a medical history which would make study agent compliance difficult or which would compromise informed consent, or recent (past 30 days) history of suicide attempts and/or current serious suicidal intention or plan as assessed by the SCID and the BDI-II;
3. currently on prescription medication that is known to interact with the study drug;
4. have current dependence on cocaine, opiates, alcohol, or benzodiazepines, as defined by DSM-IV-TR criteria;
5. have a history of alcohol dependence within the past three years;
6. have a history of mitral valve prolapse, left ventricular hypertrophy, cardiac arrhythmias, angina, myocardial infarction, acute coronary syndrome (unstable angina), cardiac syncope or presyncope, or any EKG abnormalities that suggests the presence of one of these conditions;
7. have a systolic blood pressure greater than 160, a diastolic blood pressure greater than 100 (i.e. cutoffs for stage 2 hypertension), and a heart rate greater than 70% of the maximum heart rate expected for their age (0.70(220-age)) at any of the study visits.
8. any other circumstances that, in the opinion of the investigators, would compromise participant safety;
9. have a history of sensitivity to modafinil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Shoptaw, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Vine Street Clinic, Hollywood, California, United States

REFERENCES:
- [Result] Heinzerling KG, Swanson AN, Kim S, Cederblom L, Moe A, Ling W, Shoptaw S. Randomized, double-blind, placebo-controlled trial of modafinil for the treatment of methamphetamine dependence. Drug Alcohol Depend. 2010 Jun 1;109(1-3):20-9. doi: 10.1016/j.drugalcdep.2009.11.023. Epub 2010 Jan 25. PMID 20092966
- [Result] Heinzerling KG, Shoptaw S. Gender, brain-derived neurotrophic factor Val66Met, and frequency of methamphetamine use. Gend Med. 2012 Apr;9(2):112-20. doi: 10.1016/j.genm.2012.02.005. Epub 2012 Mar 23. PMID 22445683
- [Result] Heinzerling KG, McCracken JT, Swanson AN, Ray LA, Shoptaw SJ. COMT Val158Met, BDNF Val66Met, and OPRM1 Asn40Asp and methamphetamine dependence treatment response: preliminary investigation. J Clin Psychopharmacol. 2012 Feb;32(1):135-7. doi: 10.1097/JCP.0b013e318240a48e. No abstract available. PMID 22217949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were 71 MA-dependent outpatients seeking treatment in the Los Angeles area recruitment from 4/07-9/08. Potential study participants were recruited from the community using advertisements for a study of experimental medications for MA dependence.
Pre-assignment Details: Subjects completed medical and psychiatric screening (to exclude any non-drug related Axis I disorder) and baseline assessments over a two-week/six-visit lead in.
Period: Overall Study
Arm/Group | Modafinil | Placebo
Started | 34 | 37
Completed | 14 | 13
Not Completed | 20 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil | Placebo | Total
Number analyzed (Participants) | 34 | 37 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 37 | 71
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (11.1) | 37.8 (10.1) | 38.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 25 | 25 | 50
Region of Enrollment [Number; unit: participants]
  United States | 34 | 37 | 71

OUTCOME MEASURES:

1. Primary Outcome: Clean Urine Drug Screen
Description: Urine samples, collected thrice weekly, were tested for metabolites of MA using radioimmunoassay. Each subject had a possible of 36 urine drug screens to provide during the 12 weeks of medication. An aggregate measure of urine drug screen results was calculated - the Treatment Effectiveness Score (TES) - which is the average of the sum of MA-free urine specimens provided during the treatment period by participants in each treatment condition.
Time Frame: From randomization to end of week 12
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: Clean urine drug screens
Units Other Than Participants: Urine drug screens
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 34 | 37
Number analyzed (Urine drug screens) | 590 | 564
Clean urine drug screens | 13.1 (11.5) | 12.7 (13.2)

2. Secondary Outcome: Retention
Description: The number of persons who completed the medication phase of the trial (12 weeks of medication).
Time Frame: 12 weeks
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 34 | 37
participants | 14 | 13

3. Other Pre Specified Outcome: VAS Score
Description: To measure methamphetamine craving, mean change in craving based on visual analog scale (VAS) from 0 (not at all) to 100 (extremely) from baseline to the last week of observation during the 12 week treatment period. The last observation was carried forward if not available during week 12.
Time Frame: baseline and last observation during the 12 week treatment period
Population: Intention to treat, LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 34 | 37
units on a scale | -32.5 (33.8) | -47.3 (32.6)

4. Other Pre Specified Outcome: BDI Score
Description: Self-reported depression: mean change on Beck Depression Index (BDI-II) assessed weekly during the 12 week medication phase. If the week12 measure was not available, the last observation was carried forward. 0 indicates no depression, 63 is the maximum indicating severe depression.
Time Frame: From baseline to end of treatment period (week 12).
Population: Intention to treat, LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 34 | 37
units on a scale | -11.8 (12.9) | -7 (11.2)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed at each study visit during the 12 weeks of treatment and in the follow up period (4 weeks).
Description: Subjects were questioned at each clinic visit about their general health. Any physical or clinical change or illness, whether or not considered study drug related, was recorded on the medical record chart and adverse event case report form.In case of an adverse event thought to reflect drug-related toxicity, evaluation and management ensued.
Arm/Group | Modafinil | Placebo
Serious Adverse Events (participants affected / at risk) | 3/34 | 1/37
Other Adverse Events (participants affected / at risk) | 33/34 | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modafinil (N=34) | Placebo (N=37)
Otitis media (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Not study drug related.
Acute Epididymitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Not study drug related
Injection site abscess (Infections and infestations) | 1 (1) | 0 (0) — Not study drug related
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1) — Not study drug related - MA induced
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modafinil (N=34) | Placebo (N=37)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abscess Gum (Infections and infestations) | 1 (1) | 0 (0)
Agitation (General disorders) | 1 (1) | 1 (1)
Anger (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (General disorders) | 5 (5) | 1 (1)
Aphasia (General disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back Pain (General disorders) | 1 (2) | 2 (2)
Blood Pressure Increased (Cardiac disorders) | 1 (1) | 1 (1)
Bowel Incontinena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
CHEST PAIN-L ARM (General disorders) | 1 (1) | 0 (0)
Chest tightness of (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Common Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Concentration Imparied (General disorders) | 1 (1) | 0 (0)
Congestion Nasal (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Coughing (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0)
Delusions (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (General disorders) | 2 (2) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diaphoresis (General disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (3)
Dizziness (General disorders) | 0 (0) | 1 (1)
Drowsiness (General disorders) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 1 (1) — Craving
Dry Mouth (General disorders) | 3 (3) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Earache (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ears Feel Clogged (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye Irritation (Eye disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 1 (1) | 1 (1)
Flank Pain (General disorders) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 3 (3) | 1 (1)
Fracture Bone (Social circumstances) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
GENITALIA EXTERNAL PAINFUL (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hallucitation Auditory (Psychiatric disorders) | 1 (1) | 0 (0)
Head contusion (General disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 10 (14) | 6 (10)
Hearing decreased (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Heartbeats Increased (Cardiac disorders) | 1 (2) | 2 (2)
Heartburn (Gastrointestinal disorders) | 1 (1) | 1 (1)
Herpes Simplex (General disorders) | 1 (2) | 0 (0)
Hot Flashes (General disorders) | 2 (2) | 0 (0)
Hyperactivity (General disorders) | 3 (6) | 1 (1)
Infection Upper Respiratory (Infections and infestations) | 2 (2) | 1 (1)
Insomnia (General disorders) | 10 (18) | 7 (8)
Irritability (General disorders) | 1 (1) | 2 (2)
Jitterniness (General disorders) | 4 (9) | 0 (0)
Joint Ache (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Laceration (Social circumstances) | 1 (1) | 1 (1)
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lethargy (General disorders) | 0 (0) | 1 (1)
Libido Decreased (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Light-headed (General disorders) | 2 (2) | 0 (0)
MENTAL CONCENTRATION DIFFICULTY (General disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 4 (5)
Nerve pain (General disorders) | 1 (1) | 0 (0)
Nervousness (General disorders) | 1 (1) | 0 (0)
Nightmares (General disorders) | 1 (1) | 2 (4)
Nosebleed (General disorders) | 1 (1) | 0 (0)
Pain muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Palpitation (Cardiac disorders) | 2 (2) | 0 (0)
Pneumonia (Immune system disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Rash Impetiginous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sexual Dysfunction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shakiness (General disorders) | 1 (1) | 1 (1)
Shortness of breath (General disorders) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Headache (General disorders) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sore Throat (General disorders) | 4 (4) | 0 (0)
Stomach pain (General disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tightness of chest (General disorders) | 0 (0) | 1 (1)
Tinea (Infections and infestations) | 0 (0) | 1 (1) — Ringworm
Vision Blurred (General disorders) | 1 (1) | 0 (0)
Visual disturbance (General disorders) | 0 (0) | 1 (1)
Vivid Dreams (General disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Wakefulness (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
study is powered to detect at least a moderate effect for modafinil (d = 0.50) in the overall sample; subgroups may be more meaningful

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes